CLINICAL TRIAL: NCT03156569
Title: Oral Health and Salivary Markers in Patients With Xerostomia
Brief Title: Salivary Markers in Patients With Xerostomia
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, MD DDS PhD, Universidad de Murcia
Other Study IDs: University of Murcia
Record Dates: First submitted 2017-05-01; First posted 2017-05-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland
Keywords: saliva , dental , oral health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Analysis of the saliva — IFN-, IL-10, IL-1b, IL-4 and IL-6

SUMMARY:
The purpose of this study was to investigate the salivary levels of inflammatory and their association with oral health in xerostomía patient

DETAILED DESCRIPTION:
Primary Outcome Measures:

* salivary Proinflammatory and anti-inflammatory cytokines
* questionnaire is provided to the patient for xerostomia characterization

Secondary Outcome Measures:

* Probing pocket depth
* Probing pocket depth and clinical attachment level
* Gingival index
* Plaque index
* Bleeding on probing

ELIGIBILITY:
Inclusion Criteria:

• The patient must have clinical symptoms of xerostomia (dry mouth)

Exclusion Criteria:

* Head and neck radiotherapy
* Administration anti-inflammatory drugs or antibiotic therapies within the previous 6 months
* Patients who are unable or unwilling to cooperate
* Patient suffering from cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients Oral Medicine Hospital Morales Meseguer Clinica Odontologica University
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
saliva flow rate | 2 months
  Unstimulated salivary flow rate. Pathological < or 1.5 ml/ 15 minutes.
Xerostomia | 2 months
  Visual Analogue Scale (VAS) for xerostomia severity (0 cm: no xerostomía , 10cm : very severe xerostomia ).
Interleukins | 2 months
  Analytes in saliva IFN-(pg/ml), IL-10(pg/ml), IL-1b(pg/ml), IL-4 (pg/ml)and IL-6 (pg/ml)

SECONDARY OUTCOMES:
Oral Exam | 4 months
  Caries number, natural teeth number
Periodontal evaluation | 4 months
  periodontal( gingival index, bleeding index, clinical attachment level, probing depth,number dental implant .A periodontal probe will be inserted between the tooth and the gum in the gingival sulcus and a measurement of the pocket depth will be measured by a trained dentist in all subjects according to American Academy of Periodontology classification of periodontal diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohyama K, Moriyama M, Hayashida JN, Tanaka A, Maehara T, Ieda S, Furukawa S, Ohta M, Imabayashi Y, Nakamura S. Saliva as a potential tool for diagnosis of dry mouth including Sjogren's syndrome. Oral Dis. 2015 Mar;21(2):224-31. doi: 10.1111/odi.12252. Epub 2014 May 15. PMID 24750447
- [Result] van den Berg I, Pijpe J, Vissink A. Salivary gland parameters and clinical data related to the underlying disorder in patients with persisting xerostomia. Eur J Oral Sci. 2007 Apr;115(2):97-102. doi: 10.1111/j.1600-0722.2007.00432.x. PMID 17451498
- [Result] Liukkonen J, Gursoy UK, Pussinen PJ, Suominen AL, Kononen E. Salivary Concentrations of Interleukin (IL)-1beta, IL-17A, and IL-23 Vary in Relation to Periodontal Status. J Periodontol. 2016 Dec;87(12):1484-1491. doi: 10.1902/jop.2016.160146. Epub 2016 Aug 19. PMID 27541079
- [Derived] Tvarijonaviciute A, Zamora C, Martinez-Subiela S, Tecles F, Pina F, Lopez-Jornet P. Salivary adiponectin, but not adenosine deaminase, correlates with clinical signs in women with Sjogren's syndrome: a pilot study. Clin Oral Investig. 2019 Mar;23(3):1407-1414. doi: 10.1007/s00784-018-2570-3. Epub 2018 Jul 20. PMID 30030617